CLINICAL TRIAL: NCT00239980
Title: A Phase II Randomized Study of Fragmin in Ovarian Cancer: Utility on Survival (FOCUS)
Brief Title: Fragmin in Ovarian Cancer: Utility on Survival (FOCUS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Dr. Mark Levine, Ontario Clinical Oncology Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRA6300011-FOCUS-II
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Ovarian Cancer
Keywords: antineoplastic agent; ovarian cancer; fragmin; dalteparin
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): 50 IU/kg
  Interventions: Drug: dalteparin
- B (Active Comparator): 100 IU/kg
  Interventions: Drug: dalteparin
- C (Active Comparator): 150 IU/kg
  Interventions: Drug: dalteparin

INTERVENTIONS:
Drug: dalteparin — 50, 100, 150 IU/kg administered subcutaneously once daily for 3 cycles of chemotherapy
  Other Names: brand name is fragmin

SUMMARY:
Epithelial ovarian carcinoma (EOC) is the 5th leading cause of death among women. Long-term survival is poor for the majority of women with EOC because many present with advanced disease. Chemotherapy and cytoreductive surgery produces a 50% - 60% response rate but relapse is not uncommon. Adding more systemic agents has failed to show a clear benefit in survival and is associated with unacceptable toxicity. This phase II, dose-finding, open label trial will enrol women with newly diagnosed EOC and randomize them to receive one of 3 doses of a LMWH dalteparin in conjunction with standard adjuvant taxane- and platinum-based chemotherapy. The primary outcome is disease response, measured according to Gynaecologic Cancer Intergroup (GCIG) Cancer Antigen (CA)-125 response criteria. Secondary outcomes include symptomatic venous thromboembolism, bleeding, and compliance. The dose of dalteparin associated with the best response will be tested further in a phase III randomized clinical trial in the same patient population.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to be considered for enrolment:

* Women with newly diagnosed, histologically proven EOC are potentially eligible. Patients with primary peritoneal or fallopian tube tumours of equivalent histology are also considered for enrolment. If open or true cut biopsy is not available, fine needle aspiration (FNA) showing an adenocarcinoma is considered diagnostic for EOC if all 4 (a to d) of the following conditions are satisfied:

  1. Patient has a pelvic mass, AND
  2. Any evidence of disease larger than 1 cm in the upper abdomen (unless proven stage IV), AND
  3. Normal mammography within 6 weeks of randomization, AND
  4. Serum CA-125/CEA greater than or equal to 25. If the ratio is less than 25, a barium enema (or colonoscopy) and gastroscopy (or radiological examination of the stomach) must be negative for a primary tumour.
* Between the ages of 18 and 75.
* FIGO stage IIB to IV disease.
* A pre-study CA-125 level at least twice the upper limit of normal.
* Eligible for standard adjuvant treatment with taxane- and platinum-based chemotherapy by meeting all of the following laboratory findings within 7 days prior to randomization:

  1. Absolute granulocyte count of at least 1.5 x 10 9/L (1500 per cubic millimetre).
  2. Platelet count of at least 150 x 109/L (100,000 per cubic millimetre).
  3. Serum creatinine no greater than 177 micromol/L (2.0 mg/dL).
  4. Total bilirubin level no greater than 1.5 times the upper limit of normal at the local centre.
  5. Serum alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) levels no greater than 3 times the upper limit of normal of the local centre.

Exclusion Criteria:

* Borderline ovarian tumours.
* Received prior chemotherapy or radiation therapy for EOC.
* Received mouse antibodies anytime during the 28 days prior to the pre-study CA-125 level.
* History of another malignancy, unless disease-free for 5 years or greater; non-melanomatous skin carcinoma or curatively treated carcinoma-in-situ of the cervix are excepted.
* Eastern Cooperative Oncology Group (ECOG) performance score of 3 or 4.
* Life expectancy less than 12 weeks.
* Complete bowel obstruction at the time of study enrolment.
* Receiving long-term anticoagulant therapy for an established indication (e.g., atrial fibrillation, mechanical heart valves).
* Bleeding diathesis (e.g., evidence of DIC, hereditary or acquired bleeding disorder).
* History of allergy to any heparin (e.g., heparin-induced thrombocytopenia).
* Significant cardiac history including myocardial infarction within preceding 6 months, congestive heart failure, clinically relevant atrial or ventricular arrhythmias, history of 2nd or 3rd degree heart blocks unless pacemaker is implanted.
* Serious medical conditions that preclude the administration of chemotherapy, anticoagulant therapy, or adherence to protocol, including but not exclusive to:

  1. Allergic reactions to drugs containing cremophor or compounds chemically related to taxanes or platinum analogues.
  2. Significant neurologic or psychiatric disorder that would impair obtaining informed consent and reliable follow-up.
  3. Uncontrolled hypertension despite optimal medical therapy.
  4. Active, uncontrolled infection.
* Women who are pregnant or lactating or are of childbearing potential but are not using effective contraception.
* Total body weight of less than 40 kg.
* Concurrent treatment with experimental or investigational drugs.
* Unable or unwilling to attend scheduled follow-ups.
* Unable (e.g., language barrier, mental illness) to provide informed consent.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2005-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
disease response | up to day 1 of cycle 6

SECONDARY OUTCOMES:
symptomatic venous thromboembolism | up to 7 days after last dose of dalteparin
bleeding | up to 24 hours after last dose of dalteparin
compliance | up to the end of cycle 3
death | up to the last day of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Elit, MD, Study Chair — Juravinski Cancer Centre; Agnes Lee, MD, Study Chair — Hamilton Health Sciences Henderson Division; Mark Levine, MD, Principal Investigator — McMaster University, Ontario Clinical Oncology Group; Jim Julian, MMath, Principal Investigator — McMaster University, Dept. of Clinical Epidemiology & Biostatistics
Locations (9):
- Canada (9):
  - Cross Cancer Institute, Edmonton, Alberta
  - B.C. Cancer Agency- Fraser Valley Centre, Surrey, British Columbia
  - B.C. Cancer Agency- Vancouver Centre, Vancouver, British Columbia
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Hopital Notre-Dame, Montreal, Quebec

REFERENCES:
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539